CLINICAL TRIAL: NCT02295319
Title: The Impact of Individual-based Discharges From Acute Admission Units to Home on Healthcare Utilization, Quality-of-life and Patient Experience: a Randomized Controlled Study
Brief Title: The Impact of Individual-based Discharges From Acute Admission Units to Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Discharge AAU
Record Dates: First submitted 2014-11-12; First posted 2014-11-20 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2014-11

CONDITIONS: Patient Discharge
Keywords: Discharge; Acute Admission Unit; Randomized Controlled Trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individual discharge (Experimental): Discharge based on the patients individual needs and conditions. The discharge focus on information, communication, follow-up plans and collaboration, as well as the patients understanding and accept of the discharge plan. In addition, it includes a telephone interview 2 days after discharge to home.
  Interventions: Other: Individual discharge
- Control (No Intervention): Usual discharge procedures

INTERVENTIONS:
Other: Individual discharge — See previous description in "Arms"
  Arms: Individual discharge

SUMMARY:
The present non-blinded randomized controlled trial (RCT) investigates the effect of a comprehensive discharge model in adult medical patients discharged directly home from an Acute Admission Unit (AAU). In addition, eligible patients should have, at least, one hospital admission 12 months prior to index hospitalization and be discharged for further follow-up by general practitioner, home care nursing or in an out-patient clinic. The model consists of 3 main steps during the short term stay in the AAU. First, patients are screened for pre-hospital conditions that might have contributed to the index hospitalization i.e. functional ability, ongoing treatment including drug treatment, need for additional assistance to maintain daily living, relatives, and use of e.g. hearing aid, glasses, walker. Second, at point of discharge there will be a thorough assessment of the discharge plan focusing on the patients' comprehension of the discharge plan as well as accept of the suggested treatment and follow-up. Third, within 2 days after discharge the patient will receive a discharge letter by email or postal mail written in plain language and repeating the information provided in the discharge summary to the general practitioner. Subsequently, the patient will receive a telephone follow-up from the research nurse addressing the content in the discharge letter and possible unresolved issues related to the index hospitalization. Patients in the control group receives the usual discharge practice in the AAU which does not include a discharge letter to the patient and telephone follow-up after discharge.

The primary endpoint is number of readmissions within 72 hours and 30 days after discharge. Secondary endpoints are healthcare service utilization within 30 days after discharge this includes number of contacts to general practitioner, out-of-hours physicians, emergency departments and if possible visits by home care nurses. Additionally, Quality-of-Life measured 30 days after discharge by the questionnaire EQ5D and Patient Experience of the discharge process is measured 7 days after discharge by a Danish national patient experience survey - serves as secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* medicine diagnosis
* discharged directly to home
* 1 admission during the last 12 months
* having a planned follow-up after discharge (general practitioner, home care nurse, out-patient clinic)
* read and understand Danish

Exclusion Criteria:

* demented, living outside the council of Aarhus, included in a rival study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Readmissions | 30 days

SECONDARY OUTCOMES:
Healthcare Service Utilization | 30 days
Quality of Life (EQ5D) | 30 days
Patients experience of the discharge process | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark